CLINICAL TRIAL: NCT00684554
Title: Buprenorphine Maintenance Treatment of Opioid Dependence in Primary Care: A Randomized Clinical Trial of At-Home Versus In-Office Buprenorphine Induction
Brief Title: Buprenorphine Maintenance Treatment of Opioid Dependence in Primary Care: A Randomized Clinical Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #5600; K23DA020000 (NIH)
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Opioid-Related Disorders; Heroin Dependence
Keywords: Heroin Dependence; Opioid Dependence; Primary Care; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unobserved-at home (Active Comparator): Buprenorphine Unobserved at home induction
  Interventions: Drug: Buprenorphine
- Observed (Active Comparator): Buprenorphine Observed in office induction
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Dose is determined according to the participants' individual need.
  Other Names: Bup

SUMMARY:
The study will assess the effectiveness of at-home vs. in-office induction for patients entering buprenorphine maintenance at Associates in Internal Medicine (AIM) primary care clinic.

DETAILED DESCRIPTION:
Buprenorphine maintenance is an effective treatment for opioid dependence, yet diffusion has been limited. Physician concern about induction is a reported barrier, primarily as buprenorphine may precipitate withdrawal due to its partial opioid agonist activity and high receptor binding affinity. To minimize risk, guidelines recommend in-office assessment and monitoring during induction. As this may not be feasible (e.g., time limitations), many patients are instructed to self-induct at home. While this may facilitate treatment entry, data on at-home induction are limited. The study will assess the effectiveness of at-home vs. in-office induction for patients entering buprenorphine maintenance at Associates in Internal Medicine (AIM) primary care clinic. Currently, patients receive buprenorphine maintenance at AIM as part of standard clinical practice and through an observational study (IRB 5258). Most patients are insured through Medicaid, which covers visit, medication (obtained through prescription from a local pharmacy), lab, and outside psychosocial treatment cost. In this demonstration project, 20 opioid dependent patients will be randomly assigned to at-home or in-office induction, and then monitored for 12 weeks. Ancillary psychosocial treatment will be encouraged but not required. After randomization, AIM clinic and NYSPI research visits will be scheduled weekly for 4 weeks, and then at weeks 8 and 12. The primary outcome will include a comparison of the proportion of patients successfully inducted one week after the initial primary care visit. Secondary outcomes will include: 1) Time to stabilization after buprenorphine initiation assessed by: a) Time until the patient is without withdrawal for two consecutive days, and b) Time until the patient is opioid free for two consecutive weeks; and 3) Retention-in-treatment at 4 and 12 weeks. Other secondary outcomes include patient satisfaction and change in addiction severity. These data will provide important information in buprenorphine initiation in primary care and enable determination of treatment effects size prior to future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV criteria for current opioid dependence with physical dependence and are seeking treatment
2. Recent opioid use
3. Individuals must describe opioids as their primary drug of abuse.
4. 18-65 years of age
5. Able to give informed consent and comply with study procedures
6. Financially able to receive treatment at AIM and obtain medication (e.g., Medicaid)

Exclusion Criteria:

1. DSM-IV opioid dependence without physical dependence
2. Any current Axis I psychiatric disorder(s) as defined by DSM-IV-TR that in the investigator's judgment are unstable or would be disrupted by study participation (e.g., psychosis, active suicidal or homicidal ideation).
3. Individuals who are significant risk for suicide based on their current mental state or history.
4. DSM-IV alcohol or benzodiazepine dependence with physiologic dependence.
5. Pregnancy, lactation. Women must also agree to use a method of contraception with proven efficacy and agree not to become pregnant during the study.
6. Unstable physical disorder that might make participation hazardous.
7. Individuals with a known allergy, sensitivity or adverse reaction to buprenorphine.
8. Past life-threatening idiosyncratic severe opioid withdrawal reaction (e.g., psychosis, seizure)
9. Current buprenorphine maintenance
10. Current long-acting opioid use (e.g., methadone)
11. Inability to read or understand the self-report assessment forms unaided

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik W Gunderson, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty patients were recruited between December 2007-June 2008 through referrals from clinical and research groups at Columbia University Medical Center and locally posted flyers.
Pre-assignment Details: After a structured telephone interview, participants completed in-person screening after obtaining informed consent. Of the 21 patients screened, one was excluded for active alcohol and benzodiazepine dependence.
Period: Overall Study
Arm/Group | Unobserved-at Home | Observed
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adult Opioid Dependent treatment seekers
Groups:
- Total: Total of all reporting groups
Arm/Group | Unobserved-at Home | Observed | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will Include a Comparison of the Proportion of Patients Successfully Inducted One Week After the Initial Primary Care Visit.
Description: The primary outcome will include a comparison of the proportion of patients successfully inducted one week after the initial primary care visit. Defined as in treatment, on Buprenorphine and withdrawal free.
Time Frame: one week after initial primary care visit
Population: patients who in initiated induction
Measure: Number; unit: participants
Arm/Group | Unobserved-at Home | Observed
Number analyzed (Participants) | 10 | 10
participants | 6 | 6

2. Secondary Outcome: Prolonged Withdrawal
Description: participants experiencing prolonged withdrawal beyond two days after buprenorphine induction
Time Frame: a) 2 days
Population: participants who initiated induction
Measure: Number; unit: participants
Arm/Group | Unobserved-at Home | Observed
Number analyzed (Participants) | 10 | 10
participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Unobserved-at Home | Observed
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unobserved-at Home (N=10) | Observed (N=10)
Prolonged withdrawal (Gastrointestinal disorders) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
The primary pilot study limitations are sample size and treatment setting, which restricts statistical comparison of outcomes and generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No